CLINICAL TRIAL: NCT06199622
Title: The Effect of Music on Anxiety Levels, Blood Pressure, Fetal Heart Rate and Maternal-Fetal Attachment in Pregnant Women With Gestational Hypertension
Brief Title: The Effect of Music on Pregnant Women With Gestational Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Büşra Güngör, master student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-BGUNGOR-001
Record Dates: First submitted 2023-12-06; First posted 2024-01-10 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Gestational Hypertension; Music; Blood Pressure; Anxiety; Maternal-Fetal Relations
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled intervention trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Pregnant women in the intervention group will listen to 20 minutes of music consisting of classical western music - Beethoven moonlight sonata -, classical Turkish music - Nihavend and Buselik Maqam - for three days with a MP3 player with a good sound system and headphones.
  Interventions: Other: music
- control group (No Intervention): Pregnant women in the control group did not receive 20 minutes of music for three days and routine care will continue.

INTERVENTIONS:
Other: music — 20 minutes of classical Turkish musicor classical western music
  Arms: experimental group

SUMMARY:
In this study, the effect of music on arterial blood pressure, anxiety level, fetal heart rate and maternal-fetal attachment in pregnant women with gestational hypertension will be studied and it will be conducted as a randomized controlled intervention study to examine the relationships with each other. The sample group will consist of 90 pregnant women, 45 in the intervention group and 45 in the control group. Within the scope of the study, the data will be collected using the 'Personal Information Form, State-Trait Anxiety Scale (STAI TX-I)', Maternal-Fetal Attachment Scale (MFA) created by the researcher, and the systolic blood pressure and diastolic blood pressure of each patient will be measured with a calibrated sphygmomanometer (the same sphygmomanometer was used for each patient), fetal heart rate (FHR) and fetal movements (FM) will be measured by Electronic Fetal Monitoring and Nonstress test (NST). Data will be analyzed using SPSS-25 package.

DETAILED DESCRIPTION:
In this study, the effect of music on arterial blood pressure, anxiety level, fetal heart rate and maternal-fetal attachment in pregnant women with gestational hypertension will be studied and it will be conducted as a randomized controlled intervention study to examine the relationships with each other. The sample group will consist of 90 pregnant women, 45 in the intervention group and 45 in the control group. Within the scope of the study, the data will be collected using the 'Personal Information Form, State-Trait Anxiety Scale (STAI TX-I)', Maternal-Fetal Attachment Scale (MFA) created by the researcher, and the systolic blood pressure and diastolic blood pressure of each patient will be measured with a calibrated sphygmomanometer (the same sphygmomanometer was used for each patient), fetal heart rate (FHR) and fetal movements (FM) will be measured by Electronic Fetal Monitoring and Nonstress test (NST). Data will be obtained by the researcher by face-to-face interviews with pregnant women. In addition, pregnant women in the intervention group will be given music once a day for 20 minutes at the beginning of the study. Pregnant women in the control group will continue their routine care. Data will be evaluated with SPSS-25 package.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women hospitalized with a diagnosis of Gestational Hypertension/Mild Preeclampsia (Severe Preeclamptic Pregnant Women were not included in the study),
* Pregnancy at 28 weeks of gestation and above (since NST will be performed during follow-up),
* No hearing problems (because music will be played),
* Good level of consciousness,
* Being at least literate (for consent to be obtained),
* Being over 18 years of age (for consent to be obtained),
* No communication problems,
* A live, single, healthy fetus.
* Pregnant women who verbally and in writing agreed to participate in the study

Exclusion Criteria:

* Written and verbal refusal to participate in the research,
* Illiteracy,
* Must be under 18 years of age,
* Communication problems,
* Hearing problems,
* Before the 28th week of pregnancy,
* Hospitalized for less than three days with a diagnosis of Gestational Hypertension/Preeclampsia,
* Hospitalized with a diagnosis of severe pre-eclampsia,
* Multiple pregnancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
vital signs | 6 months
  Blood pressure (mm/Hg) of pregnant women will be measured with a calibrated sphygmomanometer.
anxiety | 6 months
  Anxiety will be measured with State-Trait Anxiety Inventory (STAI TX-I) before and after the intervention. The scale consists of 20 items on a 4-point Likert scale ((1) not at all, (2) a little, (3) a lot, (4) completely). The total score value obtained can vary between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
maternal fetal attachment | 6 months
  Changes in mother-infant attachment will be measured with the Maternal-Fetal Attachment Scale (MFA) before and after the intervention. Responses are scored from 1-5, with 5 being the most positive statement. The higher the score, the higher the attachment.
Fetal heart rate | 6 months
  Nonstress test (NST) will be performed with Electronic Fetal Monitoring for an average of 20 minutes and fetal heart rate (beats per minute) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Güngör, Principal Investigator — Saglik Bilimleri Universitesi; Gülten Güvenç, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsakiridis I, Giouleka S, Arvanitaki A, Mamopoulos A, Giannakoulas G, Papazisis G, Athanasiadis A, Dagklis T. Chronic hypertension in pregnancy: synthesis of influential guidelines. J Perinat Med. 2021 Apr 20;49(7):859-872. doi: 10.1515/jpm-2021-0015. Print 2021 Sep 27. PMID 33872475
- [Background] Henderson JT, Vesco KK, Senger CA, Thomas RG, Redmond N. Aspirin Use to Prevent Preeclampsia and Related Morbidity and Mortality [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2021 Sep. Report No.: 21-05274-EF-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK574449/ PMID 34644040
- [Background] Corbijn van Willenswaard K, Lynn F, McNeill J, McQueen K, Dennis CL, Lobel M, Alderdice F. Music interventions to reduce stress and anxiety in pregnancy: a systematic review and meta-analysis. BMC Psychiatry. 2017 Jul 27;17(1):271. doi: 10.1186/s12888-017-1432-x. PMID 28750631
- [Background] Doğan, A., Akın, B., & Tanyer, D. Gebelik Döneminde Uygulanan Müzik Girişimlerinin Maternal ve Fetal Sağlığa Etkisi: Sistematik Derleme Protokolü
- [Background] Duman, M., Yüksekol, Ö. D., & Ozan, Y. D.(2021). Preeklampsili Gebelerde Gebelikle İlişkili Anksiyetenin Prenatal Bağlanmaya Etkisi. Jinekoloji-Obstetrik ve Neonatoloji Tıp Dergisi, 18(3), 907-915.).
- [Background] Purwati, Y. (2019). Blood Pressure Changes in Pregnant Women through Murratal and Classical Music Therapy. EAS Journal of Nursing and Midwifery, 1(4), 142-147
- [Background] Teckenberg-Jansson, P., Turunen, S., Pölkki, T., Lauri-Haikala, M. J., Lipsanen, J., Henelius, A., ... & Huotilainen, M. (2019). Effects of live music therapy on heart rate variability and self-reported stress and anxiety among hospitalized pregnant women: A randomized controlled trial. Nordic Journal of Music Therapy, 28(1), 7-26.
- [Background] Yüksekol, Ö. D., & Başer, M. (2020). The effect of music on arterial blood pressure and anxiety levels in pregnant women hospitalized due to mild preeclampsia: A pilot randomized controlled trial. European Journal of Integrative Medicine, 35, 101093